CLINICAL TRIAL: NCT02279888
Title: CardioMEMS HF System Post Approval Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10035
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Left-Sided Heart Failure; Congestive Heart Failure
Keywords: Pulmonary Artery Pressure Monitoring; Implantable Hemodynamic Monitor
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CardioMEMS HF System Group: Patients implanted with a CardioMEMS HF System.
  Interventions: Device: CardioMEMS HF System

INTERVENTIONS:
Device: CardioMEMS HF System — Pulmonary artery pressure sensor

SUMMARY:
The purpose of the CardioMEMS HF System Post Approval Study (PAS) is to evaluate the use of the CardioMEMS HF System in patients with NYHA class III heart failure in a commercial setting.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the safety and to report clinical performance of the CardioMEMS™ HF System in real world setting.

Prospective, non-randomized, open-label, multi-center, post-market study designed to characterize the use of the CardioMEMS™ HF System in a real-world setting in the US; N=1200. It is the condition of approval study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NYHA class III heart failure
* At least 1 heart failure hospitalization within previous 12 months
* Patients with reduced LVEF heart failure should be receiving a beta blocker for 3 months and an ACE-I or ARB for one month unless in the investigator's opinion, the patient is intolerant to beta blockers, ACE-I or ARB
* BMI ≤ 35. Patients with BMI >35 will require their chest circumference to be measured at the axillary level. If > 65 inches the patient will not be eligible for the study.
* Pulmonary artery branch diameter ≥ 7mm - (implant target artery - assessed during the right heart catheterization)

Exclusion Criteria:

* Active infection
* History of recurrent (> 1) pulmonary embolism or deep vein thrombosis
* Inability to tolerate a right heart catheterization
* A major cardiovascular event (e.g., myocardial infarction, open heart surgery, stroke, etc.) within previous 2 months
* Cardiac resynchronization device (CRT) implanted within previous 3 months
* Glomerular Filtration Rate (GFR) < 25 ml/min (obtained within 2 weeks of implant) who are non-responsive to diuretic therapy or who are on chronic renal dialysis
* Congenital heart disease or mechanical right heart valve
* Likely to undergo heart transplantation or VAD within the next 6 months
* Known coagulation disorders
* Hypersensitivity or allergy to aspirin, and/or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with NYHA class III heart failure
Sampling Method: Non-Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Stevenson, MD, Study Chair — Brigham and Women's
Locations (1):
- West Virginia Heart Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zile MR, Abraham WT, Stevenson LW, Costanzo MR, Angermann CE, Mehra MR, Desai AS, Ducharme A, Johnson N, Henderson J, Lindenfeld J. Relationship Between Remote, Ambulatory Pulmonary Artery Pressures, and All-Cause Mortality in Patients With Chronic Heart Failure. Circ Heart Fail. 2025 Jun;18(6):e012754. doi: 10.1161/CIRCHEARTFAILURE.124.012754. Epub 2025 Apr 14. PMID 40223608
- [Derived] Brinkley DM, Guglin ME, Bennett MK, Redfield MM, Abraham WT, Brett ME, Dirckx N, Adamson PB, Stevenson LW. Pulmonary Artery Pressure Monitoring Effectively Guides Management to Reduce Heart Failure Hospitalizations in Obesity. JACC Heart Fail. 2021 Nov;9(11):784-794. doi: 10.1016/j.jchf.2021.05.020. Epub 2021 Sep 8. PMID 34509410
- [Derived] DeFilippis EM, Henderson J, Axsom KM, Costanzo MR, Adamson PB, Miller AB, Brett ME, Givertz MM. Remote Hemodynamic Monitoring Equally Reduces Heart Failure Hospitalizations in Women and Men in Clinical Practice: A Sex-Specific Analysis of the CardioMEMS Post-Approval Study. Circ Heart Fail. 2021 Jun;14(6):e007892. doi: 10.1161/CIRCHEARTFAILURE.120.007892. Epub 2021 Jun 15. PMID 34129363
- [Derived] Shavelle DM, Desai AS, Abraham WT, Bourge RC, Raval N, Rathman LD, Heywood JT, Jermyn RA, Pelzel J, Jonsson OT, Costanzo MR, Henderson JD, Brett ME, Adamson PB, Stevenson LW; CardioMEMS Post-Approval Study Investigators. Lower Rates of Heart Failure and All-Cause Hospitalizations During Pulmonary Artery Pressure-Guided Therapy for Ambulatory Heart Failure: One-Year Outcomes From the CardioMEMS Post-Approval Study. Circ Heart Fail. 2020 Aug;13(8):e006863. doi: 10.1161/CIRCHEARTFAILURE.119.006863. Epub 2020 Aug 6. PMID 32757642

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients who were consented and had an attempted implant (n=1214) are included in all safety analyses. To be considered enrolled in the study, subjects must sign consent and have the CardioMEMS PA Sensor successfully implanted (n=1200).
Groups:
- CardioMEMS HF System Group: All patients who were consented and had an attempted implant (n=1214) are included in all safety analyses. To be considered enrolled in the study, subjects must sign consent and have the CardioMEMS PA Sensor successfully implanted (n=1200).
Period: Overall Study
Arm/Group | CardioMEMS HF System Group
Started | 1214
Successful Implant | 1200
6 Months Follow Up Completed | 1013
1 Year Follow Up Completed | 875
18 Months Follow Up Completed | 770
Completed | 684
Not Completed | 530
Not completed — Death | 326
Not completed — Withdrawal by Subject | 38
Not completed — Lost to Follow-up | 21
Not completed — Physician Decision | 62
Not completed — Subject Non-compliance | 43
Not completed — Not implanted | 14
Not completed — Visit not performed | 26

BASELINE CHARACTERISTICS:
Population: Patients who underwent a CardioMEMS HF System implant procedure
Groups:
- CardioMEMS HF System Group: Patients who underwent a CardioMEMS HF System implant procedure
  CardioMEMS HF System: Pulmonary artery pressure sensor
Arm/Group | CardioMEMS HF System Group
Number analyzed (Participants) | 1214
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 457
  Male | 757
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 175
  White | 1004
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 1214
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (7.9)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: % ejected] | 38.8 (17.4)

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Device and/or System Related Complication (DSRC)
Description: As defined in the study protocol, a DSRC is an adverse event that is, or is possibly, related to the device/system (wireless pressure sensor or external electronics) and has at least one of the following characteristics: is treated with invasive means (other than intramuscular medication or right heart catheterization which is used for diagnostic purposes); results in death of the subject; results in the explant of the device. The primary safety analyses were based on the following objective performance criteria: a) the lower limit of the two-sided 95% confidence interval on the freedom from DSRC rate at 24 months is greater than 80% and b) the lower limit of the two-sided 95% confidence interval on the freedom from pressure sensor failure rate at 24 months is greater than 90%. These primary safety endpoints were tested hierarchically, testing for freedom from DSRCs first, in order to control for multiplicity.
Time Frame: two years
Measure: Count of Participants; unit: Participants
Groups:
- CardioMEMS HF System Safety Group: Patients with an attempted CardioMEMS PA Sensor implant.
  CardioMEMS HF System: Pulmonary artery pressure sensor
Arm/Group | CardioMEMS HF System Safety Group
Number analyzed (Participants) | 1214
Participants | 1209
Statistical Analysis 1: Comparison: CardioMEMS HF System Safety Group; Test type: Other — the lower limit of the two-sided 95% confidence interval on the freedom from DSRC rate at 24 months is greater than 80%; p < 0.0001, t-test, 2 sided; Kaplan Meier = 0.05

2. Primary Outcome: Freedom From Pressure Sensor Failure
Description: A Sensor failure occurs when no readings can be obtained from it after troubleshooting the system to rule out any problems with the external electronics. The primary safety analyses were based on the following objective performance criteria: a) the lower limit of the two-sided 95% confidence interval on the freedom from DSRC rate at 24 months is greater than 80% and b) the lower limit of the two-sided 95% confidence interval on the freedom from pressure sensor failure rate at 24 months is greater than 90%. These primary safety endpoints were tested hierarchically, testing for freedom from DSRCs first, in order to control for multiplicity.
Time Frame: two year
Population: Subjects implanted with CardioMEMS device
Measure: Count of Participants; unit: Participants
Arm/Group | CardioMEMS HF System Group
Number analyzed (Participants) | 1200
Participants | 1199

3. Primary Outcome: Heart Failure Hospitalization (HFH) Rate
Description: Annualized HFH rate parameter at 1 year versus the HFH rate in the year prior to enrollment using an Andersen-Gill method for recurrent events and robust sandwich variances to account for within-subject correlation. If the two-sided, upper 95% confidence interval for the hazard ratio (HR) is less than 1.0, then the primary effectiveness endpoint was met.
Time Frame: one year
Population: Patients implanted with a CardioMEMS PA Sensor
Measure: Number (95% Confidence Interval); unit: hospitalization events per patient year
Arm/Group | CardioMEMS HF System Group
Number analyzed (Participants) | 1200
hospitalization events per patient year
  1 Year HFH Rate prior implant (Events per patient year) | 1.249 [1.192 to 1.308]
  1 Year HFH Rate post implant (Events per patient year) | 0.535 [0.482 to 0.594]
Statistical Analysis 1: Comparison: CardioMEMS HF System Group; Test type: Other; p < 0.0001, Andersen-Gill; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.39 to 0.47] — This analysis applies to Primary Outcome: HFH Rate

4. Other Pre Specified Outcome: Overall Survival
Description: Survival at 1 year and 24 years post-implant is reported using the Kaplan-Meier method.
Time Frame: one and two years
Measure: Number (95% Confidence Interval); unit: survival percentage
Arm/Group | CardioMEMS HF System Group
Number analyzed (Participants) | 1200
survival percentage
  Survival at 1 year post implant | 83.9 [81.7 to 85.9]
  Survival at 2 years post implant | 71.0 [68.1 to 73.6]

5. Other Pre Specified Outcome: Heart Failure Hospitalization or Death Rate
Description: The annualized HFH or death rate parameter at 1 year was compared to the HFH rate in the year prior to enrollment using an Andersen-Gill method for recurrent events and robust sandwich variances to account for within-subject correlation. If the two-sided, upper 95% confidence interval for the hazard ratio (HR) is less than 1.0, then this effectiveness endpoint was met.
Time Frame: one year
Measure: Number (95% Confidence Interval); unit: events per patient year
Arm/Group | CardioMEMS HF System Group
Number analyzed (Participants) | 1200
events per patient year
  Annualized HFH + Death 1 Year prior implant (Events per patient year) | 1.249 [1.192 to 1.308]
  Annualized HFH + Death 1 Year post implant (Events per patient year) | 0.708 [0.646 to 0.777]
Statistical Analysis 1: Comparison: CardioMEMS HF System Group; Test type: Other; p < 0.0001, Andersen-Gill; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.52 to 0.62]

6. Other Pre Specified Outcome: Patient Compliance
Description: Total daily readings divided by total number possible for daily readings as well as total weekly readings divided by total possible weekly readings
Time Frame: One and Two Years
Measure: Mean (Standard Deviation); unit: percentage of compliance
Arm/Group | CardioMEMS HF System Group
Number analyzed (Participants) | 1200
percentage of compliance
  Weekly Compliance at 1 Year | 92.8 (15.8)
  Weekly Compliance at 2 Years | 90.0 (18.2)

7. Other Pre Specified Outcome: Training Evaluation - Freedom From DRSC in Academic and Community Hospitals
Description: To assess the effectiveness of the training program, the safety and effectiveness results were analyzed for Academic Hospitals versus Community Hospitals.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Groups:
- Academic Centers Population: Subjects implanted in Academic hospitals
- Community Centers Population: Subjects implanted in Community Hospitals
Arm/Group | Academic Centers Population | Community Centers Population
Number analyzed (Participants) | 430 | 784
Participants | 428 | 781

8. Other Pre Specified Outcome: Training Evaluation - Freedom From Pressure Sensor Failure in Academic and Community Hospitals
Description: as for outcome 7
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Groups:
- Academic Centers Effectiveness Population: Subjects implanted in Academic centers
- Community Centers Effectiveness Population: Subjects successfully implanted in Community hospitals
Arm/Group | Academic Centers Effectiveness Population | Community Centers Effectiveness Population
Number analyzed (Participants) | 425 | 775
Participants | 425 | 774

9. Other Pre Specified Outcome: Training Evaluation - HF Hospitalizations Reduction in Academic and Community Hospitals
Description: as for outcome 7
Time Frame: 2 Years
Measure: Number; unit: HF hospitalizations
Arm/Group | Academic Centers Effectiveness Population | Community Centers Effectiveness Population
Number analyzed (Participants) | 425 | 775
HF hospitalizations
  HF hospitalizations one year prior implant | 588 | 1012
  HF hospitalizations one year prost implant | 245 | 383

ADVERSE EVENTS:
Time Frame: Adverse event data were collected as they occur since the subject signed the Informed consent up to 24 months follow-up, unless the patient's participation was terminated earlier.
Description: The definition in adverse events matches the clinicaltrials.gov definition
Groups:
- CardioMEMS HF System Group: Patients who underwent a CardioMEMS HF System implant
Arm/Group | CardioMEMS HF System Group
All-Cause Mortality (participants affected / at risk) | 970/1214
Serious Adverse Events (participants affected / at risk) | 970/1214
Other Adverse Events (participants affected / at risk) | 62/1214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CardioMEMS HF System Group (N=1214)
Anemia deficiencies (Blood and lymphatic system disorders) | 1 (1)
Anaemia NEC (Blood and lymphatic system disorders) | 52 (68) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Coagulopathies (Blood and lymphatic system disorders) | 1 (1)
Leukocytoses NEC (Blood and lymphatic system disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Marrow Depression and Hypoplastic Anaemias (Blood and lymphatic system disorders) | 2 (2)
Neutropenias (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenias (Blood and lymphatic system disorders) | 8 (8)
Cardiac Disorders NEC (Cardiac disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Cardiac Signs and Symptoms NEC (Cardiac disorders) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Cardiomyopathies (Cardiac disorders) | 10 (11)
Coronary Artery Disorders NEC (Cardiac disorders) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Heart Failures NEC (Cardiac disorders) | 468 (884) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 61 (68)
Mitral Valvular Disorders (Cardiac disorders) | 11 (11)
Myocardial Disorders NEC (Cardiac disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Pericardial Disorders NEC (Cardiac disorders) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Rate and Rhythm Disorders NEC (Cardiac disorders) | 23 (24) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Supraventricular Arrhythmias (Cardiac disorders) | 70 (85)
Ventricular Arrhythmias and Cardiac Arrest (Cardiac disorders) | 93 (110)
Inner Ear Signs and Symptoms (Ear and labyrinth disorders) | 3 (3)
Adrenal Cortical Hypofunctriuons (Endocrine disorders) | 1 (1)
Hyperparathyroid Disorders (Endocrine disorders) | 1 (1)
Partial Vision Loss (Eye disorders) | 1 (1)
Visual Disorders NEC (Eye disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Abdominal Hernias, site unspecified (Gastrointestinal disorders) | 2 (2)
Abdominal Wall Conditions NEC (Gastrointestinal disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Acute and Chronic Pancreatitis (Gastrointestinal disorders) | 6 (7) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Anal and Rectal Disorders NEC (Gastrointestinal disorders) | 1 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Colitis (excl infective) (Gastrointestinal disorders) | 2 (2)
Diarrhoea (excl infective) (Gastrointestinal disorders) | 8 (11)
Duodenal and Small Intestinal stenosis and obstruction (Gastrointestinal disorders) | 6 (7)
Flatulence, bloating and Distension (Gastrointestinal disorders) | 2 (2)
Gastric Ulcers and Perforation (Gastrointestinal disorders) | 3 (3)
Gastritis (excl infective) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal and Abdominal Pain (excl oral and throat) (Gastrointestinal disorders) | 31 (35)
Gastrointestinal atonic and hypomobility disorders NEC (Gastrointestinal disorders) | 3 (3) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Gastrointestinal signs and symptoms NEC (Gastrointestinal disorders) | 8 (8) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Gastrointestinal stenosis and obstruction NEC (Gastrointestinal disorders) | 9 (9) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Gastrointestinal vascular occlusion and infarction (Gastrointestinal disorders) | 2 (2)
Haemorrhoids and gastointestinal varices (excl oesophageal) (Gastrointestinal disorders) | 1 (1)
Intestinal Haemorrhages (Gastrointestinal disorders) | 1 (1)
Intestinal ulcers and perforation NEC (Gastrointestinal disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Nausea and vomiting symptoms (Gastrointestinal disorders) | 7 (9)
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 73 (91)
Oesophageal stenosis and obstruction (Gastrointestinal disorders) | 1 (1)
Oesophagitis (excl infective) (Gastrointestinal disorders) | 2 (2)
Pancreatic and retroperitoneal disorders (Gastrointestinal disorders) | 5 (8)
Pancreatic disorders NEC (Gastrointestinal disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 5 (8)
Peritoneal and retroperitoneal fibrosis and adhesions (Gastrointestinal disorders) | 1 (1)
Asthenic conditions (General disorders) | 50 (54)
Febrile disorders (General disorders) | 15 (15)
General signs and symptoms NEC (General disorders) | 9 (9) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Hernias NEC (General disorders) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Implant and catheter site reactions (General disorders) | 1 (1)
Mass conditions NEC (General disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Oedema NEC (General disorders) | 11 (16) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Pain and discomfort NEC (General disorders) | 96 (131) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Bile duct infections and inflammations (Hepatobiliary disorders) | 1 (1)
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 9 (9)
Hepatic and hepatobiliary disorders NEC (Hepatobiliary disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Hepatic failure and associated disorders (Hepatobiliary disorders) | 3 (3)
Hepatic fibrosis and cirrhosis (Hepatobiliary disorders) | 2 (2)
Hepatobiliary signs and symptoms (Hepatobiliary disorders) | 1 (1)
Allergic conditions NEC (Immune system disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Allergies to food, food additives, drugs and other chemicals (Immune system disorders) | 1 (1)
Amyloidoses (Immune system disorders) | 3 (5)
Transplant rejections (Immune system disorders) | 3 (3)
Abdominal and gastrointestinal infections (Infections and infestations) | 13 (15)
Bacterial infections NEC (Infections and infestations) | 44 (52) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Bone and join infections NEC (Infections and infestations) | 6 (6) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Breast infections (Infections and infestations) | 1 (1)
Cardiac infections (Infections and infestations) | 5 (5)
Chlostridia infections (Infections and infestations) | 10 (18)
Herpes viral infections (Infections and infestations) | 2 (2)
Infections NEC (Infections and infestations) | 25 (28) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Influenza viral infections (Infections and infestations) | 12 (12)
Klebsiella infections (Infections and infestations) | 1 (1)
Lower respiratory tract and lung infections (Infections and infestations) | 104 (135)
Pseudomonal infections (Infections and infestations) | 1 (1)
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 87 (102) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Skin structures and soft tissue infections (Infections and infestations) | 1 (1)
Upper respiratory tract infections (Infections and infestations) | 9 (10)
Urinary tract infections (Infections and infestations) | 42 (51)
Viral infections NEC (Infections and infestations) | 6 (6) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Cerebral injuries NEC (Injury, poisoning and procedural complications) | 7 (8) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Device malfunction events (Injury, poisoning and procedural complications) | 4 (4)
Device related complications (pacemaker complications) (Injury, poisoning and procedural complications) | 2 (2)
Device related complications (Injury, poisoning and procedural complications) | 7 (8)
Fractures and dislocations NEC (Injury, poisoning and procedural complications) | 10 (12) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Injuries NEC (head injury) (Injury, poisoning and procedural complications) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Limb injuries NEC (incl. traumatic amputation) (Injury, poisoning and procedural complications) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
lower limb fractures and dislocations (Injury, poisoning and procedural complications) | 1 (1)
Non-site specific injuries NEC (fall) (Injury, poisoning and procedural complications) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 38 (41) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 2 (2)
Overdoses (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fractures and dislocations (Injury, poisoning and procedural complications) | 3 (3)
Poisoning and toxicity (Injury, poisoning and procedural complications) | 1 (1)
Renal and urinary tract injuries NEC (Injury, poisoning and procedural complications) | 14 (15) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Site specific injuries NEC (Injury, poisoning and procedural complications) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Skin injuries NEC (Injury, poisoning and procedural complications) | 4 (5) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Spinal fractures and dislocations (Injury, poisoning and procedural complications) | 6 (6)
Thoracic cage fractures and dislocations (Injury, poisoning and procedural complications) | 3 (4)
Upper limb fractures and dislocations (Injury, poisoning and procedural complications) | 5 (5)
Carbohydrate tolerance analysis (incl. diabetes) (Investigations) | 1 (1)
Cardiac function diagnostic procedures (Investigations) | 3 (3)
Coagulation and bleeding analyses (Investigations) | 9 (9)
Investigations NEC (Investigations) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Liver function analyses (Investigations) | 4 (4)
Physical examination procedures (Investigations) | 3 (4)
Renal function analyses (Investigations) | 3 (3)
Therapeutic drug monitoring analyses (Investigations) | 1 (1)
Diabetes mellitus (incl. subtypes) (Metabolism and nutrition disorders) | 6 (6)
Diabetic complications NEC (Metabolism and nutrition disorders) | 1 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Electrolyte imbalance NEC (Metabolism and nutrition disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
General nutrition disorders NEC (Metabolism and nutrition disorders) | 8 (8) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Hyperglycaemic conditions NEC (Metabolism and nutrition disorders) | 14 (14) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Hypoglicaemic conditions NEC (Metabolism and nutrition disorders) | 5 (5) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Iron deficiencies (Metabolism and nutrition disorders) | 1 (1)
Magnesium metabolism disorders (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidoses (excl diabetic acidoses) (Metabolism and nutrition disorders) | 2 (2)
Potassium imbalance (Metabolism and nutrition disorders) | 37 (42)
Purine metabolism disorders NEC (Metabolism and nutrition disorders) | 10 (10) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Sodium imbalance (Metabolism and nutrition disorders) | 14 (14)
Total fluid volume decreased (Metabolism and nutrition disorders) | 33 (36)
Total fluid volume increased (Metabolism and nutrition disorders) | 32 (38)
Arthropaties NEC (Musculoskeletal and connective tissue disorders) | 3 (3) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Bursal disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint related disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 6 (8)
Muscle related signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Muscle weakness condition (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal and connective tissue signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 37 (45) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 9 (9)
Spine and neck deformities (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast and nipple neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endocrine neoplasm benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Gastric neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphomas unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Neoplasms benign site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Neoplasms malignant site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Ovarian neoplasms malignant (excl germ cell) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory tract and pleural neoplasms malignant cell type undisclosed NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 30 (35)
Central nervous system vascular disorders NEC (Nervous system disorders) | 6 (7) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Cerebellar coordination and balance disturbances (Nervous system disorders) | 1 (1)
Dementia (excl Alzheimer's type) (Nervous system disorders) | 2 (2)
Disturbances in consciousness NEC (Nervous system disorders) | 85 (98) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Encephalopaties NEC (Nervous system disorders) | 16 (17) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Encephalopaties toxic and metabolic (Nervous system disorders) | 12 (14)
Headaches NEC (Nervous system disorders) | 3 (3) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Neurological signs and symptoms (Nervous system disorders) | 22 (24)
Paralysis and paresis (excl. cranial nerve) (Nervous system disorders) | 2 (2)
Peripheral neuropathies NEC (Nervous system disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Seizures and seizure disorders NEC (Nervous system disorders) | 6 (8) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Sensory abnormalities NEC (Nervous system disorders) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Speech and languages abnormalities (Nervous system disorders) | 2 (2)
Spinal chord and nerve root disorders NEC (Nervous system disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Structural brain disorders NEC (Nervous system disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Transient cerebrovascular events (Nervous system disorders) | 10 (10)
Tremor (excl congenital) (Nervous system disorders) | 1 (1)
Device component findings (lead fracture) (Injury, poisoning and procedural complications) | 2 (2)
Device malfunctions (lead dislodgement) (Injury, poisoning and procedural complications) | 2 (2)
Non-site specific procedural complications (seroma) (Injury, poisoning and procedural complications) | 1 (1)
Device malfunction events (sensor recalibration) (Injury, poisoning and procedural complications) | 2 (2)
Implant procedure failure (Injury, poisoning and procedural complications) | 2 (2)
Non-site specific procedural complications (hematoma post-operative) (Injury, poisoning and procedural complications) | 2 (2)
Pacemaker complication (lead dislodgement) (Injury, poisoning and procedural complications) | 1 (1)
Anxiety symptoms (Psychiatric disorders) | 3 (4)
Confusion and disorientation (Psychiatric disorders) | 10 (10)
Depressive disorders (Psychiatric disorders) | 1 (2)
Mental disorders NEC (Psychiatric disorders) | 19 (21) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Substance-related disorders (Psychiatric disorders) | 1 (1)
Suicidal and self-injurious behaviour (Psychiatric disorders) | 2 (2)
Bladder and urethral symptoms (Renal and urinary disorders) | 5 (5)
Renal disorders NEC (Renal and urinary disorders) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Renal failure and impairment (Renal and urinary disorders) | 136 (166)
Renal failure complications (Renal and urinary disorders) | 4 (4)
Renal lithiasis (Renal and urinary disorders) | 2 (2)
Renal vascular and ischaemic conditions (Renal and urinary disorders) | 1 (1)
Urinary abnormalitiues (Renal and urinary disorders) | 4 (4)
Prostate and seminal vesicles infections and inflammations (Reproductive system and breast disorders) | 2 (2)
Prostatic neoplasms and hypertrophy (Reproductive system and breast disorders) | 2 (2)
Scrotal disorders NEC (Reproductive system and breast disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Vulvovaginal disorders NEC (Reproductive system and breast disorders) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 158 (215)
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 46 (66)
Conditions associated with abnormal gas exchange (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Lower respiratory tract inflammatory and immunologic conditions (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Lower respiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal disorders NEC (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Parenchymal lung disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Pleural infections and inflammations (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 15 (17) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Pulmonary hypertensions (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedemas (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Respiratory failures (excl neonatal) (Respiratory, thoracic and mediastinal disorders) | 67 (76)
Respiratory tract disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedemas (Skin and subcutaneous tissue disorders) | 3 (3)
Bullous conditions (Skin and subcutaneous tissue disorders) | 2 (2)
Dermal and epidermal conditions NEC (Skin and subcutaneous tissue disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Skin and subcutaneous tissue ulcerations (Skin and subcutaneous tissue disorders) | 4 (5)
Biliary tract and gallbladder therapeutic procedures (Surgical and medical procedures) | 1 (1)
Bladder therapeutic procedures (Surgical and medical procedures) | 1 (1)
Cardiac device therapeutic procedures (Surgical and medical procedures) | 27 (27)
Cardiac therapeutic procedures NEC (Surgical and medical procedures) | 13 (15) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Cardiac valve therapeutic procedures (Surgical and medical procedures) | 4 (4)
Gastric therapeutic procedures (Surgical and medical procedures) | 9 (9)
Hernia repairs (Surgical and medical procedures) | 3 (3)
Joint therapeutic procedures (Surgical and medical procedures) | 7 (9)
Limb therapeutic procedures (Surgical and medical procedures) | 2 (2)
Therapeutic procedures NEC (Surgical and medical procedures) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Tongue therapeutic procedures (Surgical and medical procedures) | 1 (1)
Ureteric therapeutic procedures (Surgical and medical procedures) | 1 (1)
Uterine therapeutic procedure (Surgical and medical procedures) | 1 (1)
Vascular therapeutic procedures NEC (Surgical and medical procedures) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Accelerated and malignant hypertension (Vascular disorders) | 2 (2)
Aortic aneurysm and dissections (Vascular disorders) | 4 (4)
Aortic necrosis and vascular insufficiency (Vascular disorders) | 7 (7)
Circulatory collapse an shock (Vascular disorders) | 4 (4)
Haemorrhages NEC (Vascular disorders) | 22 (25) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Non-site specific embolism and thrombosis (Vascular disorders) | 4 (5)
Non-site specific necrosis and vascular insufficiency NEC (Vascular disorders) | 3 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Non-site specific vascular disorders NEC (Vascular disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Peripheral embolism and thrombosis (Vascular disorders) | 7 (8)
Peripheral vascular disorders NEC (Vascular disorders) | 6 (8) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Peripheral vasoconstriction, necrosis and vascular insufficiency (Vascular disorders) | 6 (7)
Vascular hypertensive disorders NEC (Vascular disorders) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Vascular hypotensive disorders (Vascular disorders) | 52 (60)
Vascular injuries NEC (Vascular disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CardioMEMS HF System Group (N=1214)
Rate and rhythm disorders NEC (Cardiac disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Febrile disorders (General disorders) | 1 (1)
General signs and symptoms NEC (General disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Pain and discomfort NEC (General disorders) | 2 (2) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Allergic conditions NEC (Immune system disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Skin structures and soft tissue infections (Infections and infestations) | 1 (1)
Device malfunctions events (Injury, poisoning and procedural complications) | 14 (17)
Device related complications (Injury, poisoning and procedural complications) | 3 (3)
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Blood gas and acid base analyses (Investigations) | 1 (1)
Cardiac function diagnostic procedures (Investigations) | 5 (6)
Musculoskeletal and connective tissue signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Soft tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Device malfunctions events (sensor recalibration, repositioning, difficulty obtaining readings) (Injury, poisoning and procedural complications) | 9 (10)
Device-related complications (migration of implant) (Injury, poisoning and procedural complications) | 5 (5)
Non-site specific procedural complications (hematoma, bleeding, incision site complications) (Injury, poisoning and procedural complications) | 5 (5)
Non-site specific injuries NEC (wound) (Injury, poisoning and procedural complications) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Skin injuries NEC (bruising) (Injury, poisoning and procedural complications) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Renal failure and impairment (Renal and urinary disorders) | 1 (1)
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Therapeutic procedures NEC (Surgical and medical procedures) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Vascular therapeutic procedures NEC (Surgical and medical procedures) | 1 (1) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.
Haemorrhages NEC (Vascular disorders) | 4 (4) — Not Elsewhere Classifiable (NEC) is used in a MedDRA code description that indicates that a more specific category is not provided in the tabular list of codes and no amount of additional information will alter the code.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT02279888/Prot_SAP_ICF_000.pdf